CLINICAL TRIAL: NCT05156762
Title: Optimizing the Body Mass Index: A Randomized Clinical Trial to Assess the Efficacy of Bariatric Surgery vs Medical Weight Loss in Morbidly Obese Patients Prior to Total Joint Arthroplasty
Brief Title: Total Joint Arthroplasty (TJA) Weight Loss Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was halted prematurely due to a lack of resources to support the study.
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-41295
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Osteoarthritis, Hip; Osteoarthritis, Knee; Obesity, Morbid
Keywords: Bariatric surgery; Medical weight loss; Total Hip Arthroplasty (THA); Total Knee Arthroplasty (TKA); Total Joint Arthroplasty (TJA); Body Mass Index >40 kg/m2; Prosthetic Joint Infection
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee; Obesity, Morbid | interventions — Bariatric Surgery; Arthroplasty, Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bariatric surgery group (Experimental): Participants randomized to the bariatric surgery arm will undergo either a laparoscopic sleeve gastrectomy or a laparoscopic gastric bypass to achieve a BMI ≤ 40 kg/m2.
  Interventions: Procedure: Bariatric surgery; Other: Patient research surveys; Procedure: Total joint arthroplasty (TJA)
- Medical weight loss group (Experimental): Participants randomized to the medical weight loss study arm will attempt to lose weight through diet, exercise, and potentially pharmacotherapy an effort to lower their BMI to ≤ 40 kg/m2.
  Interventions: Behavioral: Medical weight loss; Other: Patient research surveys; Procedure: Total joint arthroplasty (TJA)
- "Usual Standard of Care" (Other): Patients randomized to the "usual standard of care" study arm will be counseled on the importance of losing weight to optimize their BMI and will be provided with referral information (name and clinic number) to either the bariatric surgery or medical weight loss clinics.
  Interventions: Procedure: Total joint arthroplasty (TJA); Other: Usual standard of care

INTERVENTIONS:
Procedure: Bariatric surgery — Patients randomized to the bariatric surgery study arm will undergo either a laparoscopic sleeve gastrectomy or a laparoscopic gastric bypass - this decision would be a joint decision made between the study participant and the bariatric surgeon after consideration of the patient's overall goals with weight loss and discussion of the risks and benefits of each procedure.
  Arms: Bariatric surgery group
Behavioral: Medical weight loss — Study participants randomized to the medical weight loss study arm will have consultations with nutritionists, dieticians, and endocrinologists, and will make dietary and lifestyle changes in an effort to lower their BMI to ≤ 40 kg/m2. Patients may also be placed on pharmacotherapy to assist with weight loss.
  Arms: Medical weight loss group
Other: Patient research surveys — Patients will have a telemedicine visit every 3 months with an orthopaedic surgery physician assistant to review their latest BMI and to complete a patient research survey to assess the patient's feelings regarding their progress. The telemedicine visits every 3 months are unique to the clinical trial and these visits would not otherwise occur if the patient was not enrolled in the trial. If patients are found to not be advancing toward the BMI goal of ≤ 40 kg/m2, these patient research surveys can be used to make individualized adjustments, based on recommendations from dieticians and the medical nutritionist.
  Arms: Bariatric surgery group; Medical weight loss group
Procedure: Total joint arthroplasty (TJA) — Once the study participant meets the target BMI goal of ≤ 40 kg/m2, they will undergo TJA. Patients will be followed for 2 years after undergoing TJA.
Other: Usual standard of care — Patients randomized to the "usual standard of care" study arm will be counseled on the importance of losing weight to optimize their BMI and will be provided with referral information (name and clinic number) to either the bariatric surgery or medical weight loss clinics. They will be urged to make an appointment or to seek any other interventions they choose to help lower their BMI, but no appointments will be made for them. A follow up visit in 6 months and 1 year will be made for them in the arthroplasty clinic to reassess their progress. Referral information will again be provided at 6 months if no progress has been made.
  Arms: "Usual Standard of Care"

SUMMARY:
This is a randomized clinical trial (RCT) to assess the efficacy of bariatric surgery vs medical weight loss vs. the "usual standard of care" to optimize a morbidly obese patient with end-stage osteoarthritis of the hip or knee joint for total joint arthroplasty (TJA).

The study population will include patients with hip or knee joint osteoarthritis and BMI (Body Mass Index) > 40 kg/m2 who are evaluated in the joint arthroplasty clinic at Boston Medical Center.

The primary objective of the study is to determine if bariatric surgery or medical weight loss is more effective than the usual standard of care in optimizing a morbidly obese patient with osteoarthritis of the hip or knee joint for TJA. This will be determined by comparing the number of patients within each group who are able to lose weight through either bariatric surgery, medical weight loss, or the usual standard of care to achieve a BMI ≤ 40 kg/m2 to eventually undergo TJA.

The secondary objectives of this study are to compare total operative time, postoperative complication rates, readmission rates, percentage of total body weight lost, revision rate, and reoperation rate. The ability of patients within each study arm to maintain a BMI ≤ 40 kg/m2 for up to 2 years after undergoing TJA will also be assessed, as well as their level of satisfaction before and after being in the study.

DETAILED DESCRIPTION:
In this prospective RCT, eligible participants will be randomized to one of three arms - the bariatric surgery study arm, the medical weight loss study arm, or the "usual standard of care" study arm. Each patient's progress will be monitored during visits by study personnel. Participants will also have telemedicine visits with an arthroplasty physician assistant every 3 months to ensure they are making progress in terms of weight loss and becoming a safer candidate for TJA. Participants will complete research surveys every 3 months during the telemedicine visits to provide feedback regarding their progress and weight loss methods.

After the study participant has achieved a BMI ≤ 40 kg/m2, they will undergo TJA and will be seen postoperatively in the arthroplasty clinic for routine follow up visits. Patients will continue to complete patient research surveys every 3 months via telemedicine for up to 2 years to provide feedback regarding how they are managing with their weight loss after undergoing TJA.

ELIGIBILITY:
Inclusion criteria:

* Patient must be 18 years or older who has met the clinical/standard care criteria for TJA (patient must have exhausted conservative measures to treat hip or knee joint arthritis (NSAIDS, physical therapy, corticosteroid injections)), except patient has a BMI > 40 kg/m2
* Patient must be interested in TJA as a treatment option
* Patient must be willing to be randomized to either a bariatric surgery study arm, a medical weight loss study arm, or a "usual standard of care" study arm

Exclusion Criteria:

* Patient has undergone prior laparoscopic sleeve gastrectomy or gastric bypass
* Patient has undergone prior hip or knee joint replacement for the affected joint
* Active substance use disorder
* Females with child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2025-09-07 (Actual); Study Completion 2025-09-07 (Actual)

PRIMARY OUTCOMES:
Bariatric surgery to achieve a BMI ≤ 40 kg/m2 | 12 months
  The number of patients who are able to achieve a BMI ≤ 40 kg/m2 prior to total joint arthroplasty (TJA) will be analyzed.
Medical weight loss to achieve a BMI ≤ 40 kg/m2 | 12 months
  The number of patients who are able to achieve a BMI ≤ 40 kg/m2 prior to total joint arthroplasty (TJA) will be analyzed.

SECONDARY OUTCOMES:
Percentage change in body weight | Baseline, day of TJA
  The percentage change in body weight lost will be calculated from baseline to TJA
Total TJA operative time | Day of surgery
  The total number of minutes will be abstracted from the operative report
Length of hospital stay for TJA procedure | Day of surgery until discharge from hospital, up to 7 days
  The total number of days will be abstracted from the electronic health record (EHR).
Surgical site infection rate | 90 days after TJA
  The proportion of participants who develop a postoperative surgical site infection
Venous thromboembolism rate | 90 days after TJA
  The proportion of participants who develop a postoperative deep venous thrombosis
Hematoma rate | 90 days after TJA
  The proportion of participants who develop a postoperative hematoma
Urinary tract infection rate | 90 days after TJA
  The proportion of participants who develop a postoperative urinary tract infection
Cardiac event rate | 90 days after TJA
  The proportion of participants who have a postoperative cardiac event
Prosthetic joint infection rate | 90 days after TJA
  The proportion of participants who have a postoperative prosthetic joint infection
90 day postoperative readmission rate | 90 days after TJA
  The rate of hospital readmission 90 days after TJA
24 month revision rate | 24 months
  Need for total hip or total knee arthroplasty component revision after primary total hip or total knee arthroplasty
24 month reoperation rate | 24 months
  Need for reoperation for reasons other than component failure (surgical site infection, tendon injury) after primary total hip or total knee arthroplasty
Maintained a BMI ≤ 40 kg/m2 post TJA | 24 months post TJA
  The number of participants who maintained a BMI ≤ 40 kg/m2 for 24 months
Change in patient satisfaction with weight loss procedure | Baseline, 24 months
  An investigator developed questionnaire will ask a question about how satisfied participants are with the weight loss procedure used from very satisfied to not at all satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: David M Freccero, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No